CLINICAL TRIAL: NCT07329075
Title: Design and Development of a Soft Robotic Glove for Enhanced Task-Oriented Training in Stroke Rehabilitation: Incorporating Dual-Chamber Actuators and Flexible Magnetoelastic Force Sensors
Brief Title: Soft Robot for Rehabilitation of Hand Function After Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Raymond KY Tong, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2023.657
Record Dates: First submitted 2025-12-29; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Stroke
Keywords: upper limb; stroke rehabilitation; soft robotics
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- new soft robotic glove (Experimental): which allows the pressure of the dual-chamber actuators to achieve full DOF for the thumb and fingers
  Interventions: Device: new soft robotic glove
- new soft robotic glove control (Active Comparator): providing only flexion and extension like most robotic systems in the clinical setting
  Interventions: Device: new soft robotic glove
- regular rehabilitation control (No Intervention): Participants will follow their own regular rehabilitation program.

INTERVENTIONS:
Device: new soft robotic glove — a soft robotic glove, with dual-chamber actuators
  Arms: new soft robotic glove; new soft robotic glove control

SUMMARY:
The goal of this clinical trial is to investigate the feasibility of using the Soft Forearm Robot system for wrist and forearm recovery of hemiplegic subjects suffered from stroke.

Participant will attend 20 training sessions and 3 assessment sessions. This system will leverage electromyography (EMG) signals for intention detection and regulating the movement and the contact for different tasks and objects, ensuring adaptive and precise control for rehabilitation tasks. A systematic clinical study involving sixty stroke patients divided into three groups will evaluate the effectiveness of our innovative design compared to conventional rehabilitation methods. By conducting a randomized controlled trial (RCT), we aim to provide robust evidence on the benefits of our advanced robotic glove design in stroke rehabilitation. We hope our work will significantly advance the field of rehabilitation robotics by improving therapeutic practices, enhancing recovery outcomes, and elevating the quality of life for those facing hand mobility challenges. By integrating new soft robotic hand design with practical application, we aim to create an effective rehabilitation solution for everyone who needs it.

ELIGIBILITY:
Inclusion Criteria:

* chronic stage (6 months post-onset);
* adequate cognition to follow study instructions;
* being able to sit for 30 minutes;
* having detectable residual EMG signals from the affected side's flexor digitorum (FD) and extensor digitorum (ED) muscles, as well as the abductor pollicis brevis (APB) and flexor pollicis longus (FPL); and
* Modified Ashworth Scale (MAS) score indicating levels of finger spasticity of 0, 1, 1+, 2, and 3 (i.e., 0 = no muscle tone to 3 = increase in tone, difficult in passive movement).

Exclusion Criteria:

* severe dysphasia,
* conditions that could hinder study compliance, and
* certain medical or psychological disorders, such as alcoholism and substance abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment for Upper Extremity (FMA-UE) | 3-month after intervention
  It is used to evaluate and measure upper-limb recovery in post-stroke hemiplegic patients, and items are scored on a 3-point ordinal scale

SECONDARY OUTCOMES:
Action Research Arm Test (ARAT) | 3-month after intervention
  The ARAT is a 19-item measure divided into 4 sub-tests (grasp, grip, pinch, and gross arm movement) to assess upper limb functioning
Modified Ashworth Scale (MAS) | 3-month after intervention
  It measures the spasticity level of wrist, elbow and finger joint.
Box and Block Test (BBT) | 3-month after intervention
Maximum Grip Strength (GRS) | 3-month after intervention
active range of motion (AROM) of fingers | 3-month after intervention
  range of motion is a measurement to identify how far the person's joints range can move in flexion/extension
5Q-5D-5L questionnaire | 3-month after intervention
  It is a quality of life questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Tong, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Department of Biomedical Engineering, The Chinese University of Hong Kong, Hong Kong, Hong Kong